CLINICAL TRIAL: NCT07319962
Title: Investigation of Arterial Stiffness, Intercostal Muscle Oxygenation, Aerobic and Anaerobic Exercise Capacity in Elite American Football Players
Brief Title: Arterial Stiffness Intercostal Muscle Oxygenation and Aerobic-Anaerobic Capacity in Elite American Football Players
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi2708
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Arterial Stiffness; Football Players; Muscle Oxygenation
Keywords: American football; arterial stiffness; muscle oxygenation; aerobic capacity; anaerobic capacity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elite male American football players: Demographic characteristics were recorded. Inclusion criteria for the elite American football group were being a male athlete aged 18-30 years and volunteering to participate. Exclusion criteria included having any acute infection, orthopedic, neurological, or sensory problems (hearing, vision, or cooperation difficulties) that could interfere with measurements, a history of smoking, alcohol consumption, or COVID-19 infection, and use of medications or antioxidant supplements. Aerobic exercise capacity was evaluated using the Incremental Shuttle Walking Test (ISWT), anaerobic exercise capacity with the Vertical Jump Test, arterial stiffness using the SphygmoCor® XCEL Pulse Wave Analysis (PWA) Arteriograph, and intercostal muscle oxygenation by the Moxy® Muscle Oxygen Monitor.
- Health Controls: Demographic characteristics were recorded. The sedentary group (sedentary individuals were defined as those engaging in less than 150 minutes per week of moderate-intensity physical activity or its equivalent, according to WHO guidelines, inclusion criteria were being a male aged 18-30 years and volunteering to participate, while exclusion criteria included any acute, orthopedic, neurological, or sensory condition that might interfere with the assessments, as well as having a regular exercise habit. Aerobic exercise capacity was evaluated using Incremental Shuttle Walking Test (ISWT), anaerobic exercise capacity with the Vertical Jump Test, arterial stiffness using the SphygmoCor® XCEL Pulse Wave Analysis (PWA) Arteriograph, and intercostal muscle oxygenation by the Moxy® Muscle Oxygen Monitor.

SUMMARY:
American football has become an increasingly popular sport in Türkiye, and one of the key determinants of success in this discipline is the development of strong aerobic and anaerobic exercise capacities. Previous research has examined arterial stiffness in various athletic populations, including endurance athletes, wrestlers, badminton players, volleyball players, and soccer players. These studies highlight the importance of detailed cardiovascular and hemodynamic evaluation to identify potential risk groups and to better understand sport-specific physiological adaptations. In sports requiring prolonged physical effort, maximal oxygen uptake is a major determinant of performance, underscoring the need to assess this parameter in elite athletic populations. Although a limited number of studies have investigated aerobic and anaerobic exercise capacities in American football athletes, no research to date has evaluated arterial stiffness or intercostal muscle oxygenation in this group.

The present study aims to investigate arterial stiffness, intercostal muscle oxygenation, aerobic and anaerobic exercise capacity, and upper-extremity endurance in elite American football players compared with sedentary individuals. A cross-sectional study design will be used. Elite male athletes from the Gazi University American Football Team who volunteer to participate will be included, and their results will be compared with age- and sex-matched sedentary individuals. A total of 15 elite male athletes and 15 sedentary participants aged 18-30 years will be enrolled. All participants will undergo standardized assessments of arterial stiffness, intercostal muscle oxygenation, aerobic and anaerobic capacity, and upper-extremity endurance.

Normality of variables will be assessed using visual inspection and the Kolmogorov-Smirnov and Shapiro-Wilk tests. Descriptive statistics will be reported as means, standard deviations, and 95% confidence intervals for normally distributed variables, and medians with interquartile ranges (25th-75th percentiles) for non-normally distributed variables. Frequencies and percentages will be used for categorical data. Between-group comparisons will be conducted using the independent samples t-test for normally distributed variables and the Mann-Whitney U test for non-normally distributed variables. Categorical variables will be analyzed using the chi-square test. A p-value of <0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
American football is a sport that demands strength, speed, courage, teamwork, and tactical intelligence, and is played with three units-offense, defense, and special teams-over four quarters of 15 minutes each. Beyond technical and tactical training, aerobic and anaerobic power, speed, endurance, body composition, flexibility, coordination, and motor skills are fundamental contributors to performance. From a mechanical perspective, American football is classified as a moderate-dynamic, moderate-static sport, while metabolically it is predominantly anaerobic. Regular physical training plays a critical role in both the prevention and management of cardiovascular disease. Arterial stiffness is an established biomarker of vascular health and an independent determinant of cardiovascular risk. Although the term refers broadly to reduced elasticity, increased rigidity, or diminished distensibility of the arterial wall, all reflect impaired vascular compliance. Progressive arterial stiffening fosters a vicious cycle: rising aortic pressure accelerates vascular damage, promotes left ventricular hypertrophy, increases myocardial oxygen demand, and disrupts diastolic function. Research examining aortic impedance suggests that age-related increases in arterial stiffness occur more slowly in individuals who engage in lifelong regular exercise, although changes that emerge later in life may be irreversible.

Acute aerobic exercise has been shown to transiently improve arterial compliance, with increases of up to 30-40%, returning to baseline approximately one hour after exercise due to enhanced vasodilation. Studies evaluating athletes' brachial and central blood pressure and pulse wave velocity indicate that high-performance sport does not adversely affect arterial stiffness, and proposed reference values may support more detailed cardiovascular and hemodynamic assessment in elite athletic populations. Notably, no studies have specifically examined arterial stiffness in elite American football players. Based on existing evidence, it is anticipated that these athletes will exhibit lower arterial stiffness than sedentary individuals, suggesting reduced cardiovascular risk-a finding that may help identify at-risk groups more accurately.

Assessment of muscle oxygen metabolism in athletes is also crucial. During high-intensity competition, increased ventilatory demand can reduce blood flow to locomotor muscles, contributing to exercise intolerance and premature fatigue. Intercostal muscle oxygenation has been shown to be closely associated with peak oxygen uptake in athletes. As ventilation increases, the metabolic cost of breathing and oxygen consumption rise, elevating the respiratory muscles' oxygen requirements. The ability to adequately deliver oxygen to these muscles is therefore functionally important and merits investigation. However, no studies to date have evaluated intercostal muscle oxygenation in American football players.

Although several studies have explored physical and physiological characteristics across various sports, research specifically examining athletes engaged in American football-particularly in Türkiye, where the sport is expanding at the university level-remains limited. In prolonged athletic activity, maximal oxygen uptake (VO₂max) is a critical determinant of performance, reflecting the capacity to transport oxygen from inspired air to skeletal muscle mitochondria. At exercise intensities beyond the point at which cardiac output plateaus, the respiratory system must work disproportionately harder to maintain oxygen delivery to active tissues. VO₂max fundamentally represents the oxidative capacity of skeletal muscle mitochondria; higher values support the ability to sustain exercise for longer durations under stable physiological conditions. Aerobic capacity therefore depends on the integrated function of pulmonary, cardiovascular, hematologic, and muscular oxidative systems.

Anaerobic performance also plays a key role in sports requiring high-intensity, short-duration exertion. Energy for such activities is provided primarily through phosphagen and glycolytic pathways, which generate ATP rapidly but in limited quantities, whereas aerobic metabolism produces ATP at a slower rate but with virtually unlimited capacity. The phosphagen system supports explosive movements lasting up to approximately 15 seconds; activities lasting 15-30 seconds rely on both phosphagen and glycolytic pathways; and efforts of around 30 seconds depend almost entirely on glycolysis. Anaerobic performance varies according to individual and environmental factors, but regular training enhances these systems significantly. Athletes with higher anaerobic capacities typically exhibit greater fast-twitch muscle fiber content, larger muscle cross-sectional area, and superior muscle strength-factors that contribute to essential performance attributes such as sprinting and explosive lower-limb force.

Despite the central role of these physiological determinants, no research has examined arterial stiffness in elite American football players, and studies evaluating intercostal muscle oxygenation as well as aerobic and anaerobic capacities in this population are scarce. Therefore, the present study aims to evaluate arterial stiffness, intercostal muscle oxygenation, and aerobic and anaerobic exercise capacity in elite American football players and to compare these outcomes with those of sedentary individuals.

ELIGIBILITY:
Inclusion criteria for the elite American football group :

* Being a male athlete aged 18-30 years
* Volunteering to participate

Exclusion criteria for the elite American football group:

* Having any acute infection, orthopedic, neurological, or sensory problems (hearing, vision, or cooperation difficulties) that could interfere with measurements
* A history of smoking
* A history of alcohol consumption
* A history of COVID-19 infection
* Use of medications or antioxidant supplements

Inclusion criteria for the sedentary group

* Being a male aged 18-30 years
* Volunteering to participate

Exclusion criteria for the sedentary group

* Included any acute, orthopedic, neurological, or sensory condition that might interfere with the assessments
* Having a regular exercise habit

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty participants, including 15 American football players and 15 healthy controls, were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | First Day
  Arterial stiffness was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters. The device provided measures of aortic systolic blood pressure (SBP), aortic pulse pressure (APP), augmentation pressure (AP), augmentation index (AIx), heart rate-corrected augmentation index (AIx@75), aortic diastolic pressure (DBP), mean arterial pressure (MAP), heart rate (HR), and ejection duration (ED).
Aortic systolic blood pressure (SBP) | First Day
  Aortic systolic blood pressure (SBP) was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Aortic pulse pressure (APP) | First Day
  Aortic pulse pressure (APP)was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Augmentation pressure (AP) | First Day
  Augmentation pressure (AP) was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Heart rate-corrected augmentation index (AIx@75) | First Day
  Heart rate-corrected augmentation index (AIx@75) was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Aortic diastolic pressure (DBP) | First Day
  Aortic diastolic pressure (DBP) was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Mean arterial pressure (MAP) | First Day
  Arterial stiffness was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Heart rate (HR) | First Day
  Heart rate (HR) was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Ejection duration (ED) | First Day
  Ejection duration (ED) was assessed noninvasively using the SphygmoCor XCEL® system (AtCor Medical, Sydney, Australia), a device with established validity and reliability for evaluating central hemodynamic parameters.
Muscle oxygenation | First Day
  Muscle oxygenation was assessed using the Moxy® Monitor (Fortiori Design LLC, Minnesota, USA), a small, lightweight, and wireless near-infrared spectroscopy (NIRS) device that measures local muscle oxygen saturation (SmO₂) and total hemoglobin (THb) in the capillary bed of the underlying muscle tissue.
Aerobic exercise capacity | First day
  Maximal exercise capacity was evaluated using the ISWT, a standardized, externally paced, symptom-limited field test that progressively increases walking speed at one-minute intervals.

SECONDARY OUTCOMES:
Anaerobic exercise capacity | First day
  Anaerobic capacity was assessed using the Vertical Jump Test (VJT), a valid and practical field-based method for evaluating lower-limb power and anaerobic performance. The test was performed on a flat, non-slip surface under standardized conditions. Participants stood upright with feet shoulder-width apart and arms fully extended overhead to determine standing reach height. Subsequently, a maximal countermovement jump was performed by rapidly flexing the knees and explosively extending the lower extremities, without using the arms for assistance. Jump reach height was recorded, and vertical jump height was calculated as the difference between standing reach and jump reach. The test was repeated 3-5 times with adequate rest between trials to minimize fatigue, and the highest jump was used for analysis.
Anaerobic power | First day
  Anaerobic power was assessed using a vertical jump test and calculated with a validated formula based on jump height and body mass. Participants performed maximal countermovement vertical jumps following a standardized warm-up. Hands were kept on the hips to minimize upper-extremity contribution. Jump height was measured using a validated system, and the highest value obtained was used for analysis. Anaerobic power (W) was calculated as √(4.9 × body mass [kg]) × √(jump height [m]). This method provides an indirect but reliable estimation of lower-extremity anaerobic power and reflects the ability to generate high power output during short-duration explosive movements.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yoleri, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, Prof, Study Director — Gazi University; Neslişah Tunçay, Pt, Principal Investigator — Gazi University; Aleyna Gökdeniz, Pt, Principal Investigator — Gazi University; Bünyamin Ertuş, Pt, Principal Investigator — Gazi University; Esin Yağmur Kart, Pt, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Cardiopulmonary Physiotherapy and Rehabilitation, Ankara, Çankaya 06490, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ross A, Leveritt M. Long-term metabolic and skeletal muscle adaptations to short-sprint training: implications for sprint training and tapering. Sports Med. 2001;31(15):1063-82. doi: 10.2165/00007256-200131150-00003. PMID 11735686
- [Result] Mayorga-Vega D, Aguilar-Soto P, Viciana J. Criterion-Related Validity of the 20-M Shuttle Run Test for Estimating Cardiorespiratory Fitness: A Meta-Analysis. J Sports Sci Med. 2015 Aug 11;14(3):536-47. eCollection 2015 Sep. PMID 26336340
- [Result] Allen TW, Vogel RA, Lincoln AE, Dunn RE, Tucker AM. Body size, body composition, and cardiovascular disease risk factors in NFL players. Phys Sportsmed. 2010 Apr;38(1):21-7. doi: 10.3810/psm.2010.04.1758. PMID 20424398
- [Result] Bangsbo J, Mohr M, Krustrup P. Physical and metabolic demands of training and match-play in the elite football player. J Sports Sci. 2006 Jul;24(7):665-74. doi: 10.1080/02640410500482529. PMID 16766496
- [Result] Perrey S, Quaresima V, Ferrari M. Muscle Oximetry in Sports Science: An Updated Systematic Review. Sports Med. 2024 Apr;54(4):975-996. doi: 10.1007/s40279-023-01987-x. Epub 2024 Feb 12. PMID 38345731
- [Result] Ashor AW, Lara J, Siervo M, Celis-Morales C, Mathers JC. Effects of exercise modalities on arterial stiffness and wave reflection: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Oct 15;9(10):e110034. doi: 10.1371/journal.pone.0110034. eCollection 2014. PMID 25333969
- [Result] Kresnajati S, Lin YY, Mundel T, Bernard JR, Lin HF, Liao YH. Changes in Arterial Stiffness in Response to Various Types of Exercise Modalities: A Narrative Review on Physiological and Endothelial Senescence Perspectives. Cells. 2022 Nov 9;11(22):3544. doi: 10.3390/cells11223544. PMID 36428973